CLINICAL TRIAL: NCT05750758
Title: A Randomized Controlled Trial of Rivaroxaban Combined With Dual Antiplatelet Therapy Versus Dual Antiplatelet Therapy Alone 1 Month After Drug-coated Balloon Angioplasty in Patients With Acute Coronary Syndrome Without High Bleeding Risk
Brief Title: Rivaroxaban Combined With DAPT Versus DAPT Alone After Drug-coated Balloon Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HenanICE202203
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAPT+rivaroxaban (Experimental): Rivaroxaban 2.5 mg bid + aspirin 100 mg qd + ticagrelor 90 mg bid was used for 1 month after operation, and then aspirin 100 mg + ticagrelor 90 mg bid was used for 5 months.
  Interventions: Drug: rivaroxaban
- DAPT (No Intervention): aspirin 100 mg qd + ticagrelor 90 mg bid for 6 months.

INTERVENTIONS:
Drug: rivaroxaban — rivaroxaban 2.5mg bid for 1m
  Arms: DAPT+rivaroxaban

SUMMARY:
The target population of this interventional study was ACS patients with drug-coated balloons. The main discussion : 1.1 months of rivaroxaban combined with dual antiplatelet therapy compared with dual antiplatelet therapy alone, late lumen loss at 6 months. 2. To determine the safety of the regimen with bleeding events as the end point. Subjects were randomly assigned to two groups, one receiving routine DAPT for six months and one receiving DAPT plus one month of rivaroxaban 2.5 mg bid

DETAILED DESCRIPTION:
Drug-coated balloon ( DCB ) is to apply anti-intimal hyperplasia drugs to the surface of the balloon. When the balloon reaches the diseased blood vessel and is stretched and expanded, it contacts the intima of the blood vessel wall. By tearing the intima of the blood vessel and pressing, the transfer drug is quickly released to the intima of the blood vessel, thereby preventing restenosis after vascular intervention. Pretreatment is a key step in the use of drug balloons in situ macroangiopathy. At present, it is required that the residual stenosis of the lesion during pretreatment is ≤ 30 %, and there is no distal blood flow restrictive dissection and hematoma. The relationship between dissection hematoma and residual stenosis is difficult to deal with. Some small dissections are beneficial to the absorption of DCB anti-proliferative drugs by the vascular wall. The larger dissection may cause the thrombus to persist in the vascular wall, resulting in late lumen loss after organization. Rivaroxaban is a new oral anticoagulant, which is gradually used in the treatment of coronary heart disease. At present, there is no clinical study on the prognosis of vascular dissection in DCB. Based on the above research background, we designed the following trial, aimed to study in ACS population, vascular lumen access + hemorrhagic events as the end point, try to clear 1 month rivaroxaban combined with dual antiplatelet therapy compared with single dual antiplatelet therapy effect.

ELIGIBILITY:
Inclusion Criteria:

* ACS patients who meet the indications of percutaneous coronary intervention
* The reference diameter of the target vessel was ≥2.75mm
* Target lesions were treated with a drug-coated balloon catheter (DCB) for PCI
* According to IVUS assessment, the target lesions were dissected and accumulated medium without affecting distal blood flow

Exclusion Criteria:

* <18 or >60 years old
* Bridging vessels or stent restenosis
* Unable to sign written informed consent
* Female patients during pregnancy or lactation (for women who have not stopped menstruation, pregnancy test should be performed within 7 days prior to enrollment in this study)
* Antiplatelet agents and anticoagulants are not available; Have heparin, contrast agent and other allergies
* The subjects were participating in other uncompleted clinical trials
* Scheduled elective surgery
* Life expectancy is less than 1 year
* Patients with high blood risk
* Has long-term oral anticoagulant therapy adaptation
* Cardiogenic shock
* Patients with severe intraoperative dissection or hematoma requiring stent rescue

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
late lumen loss ( LLL) | 6 months
  Evaluation of postoperative target vessel LLL at follow-up using QCA

SECONDARY OUTCOMES:
Vascular dissection healing | 6 months
  Re-use CAG to evaluate the vascular reexamination of the original dissection
Minimum lumen area | 6 months
  using CAG
Cardiovascular death | 6 months
  All deaths are counted as cardiovascular deaths unless there is a clear determination of other causes
Target vessel myocardial infarction | 6 months
  CAG confirms
Clinical-driven revascularization of target lesions | 6 months
  Clinical-driven revascularization of target lesions
Bleeding events defined by BARC | 6 months
  Bleeding events defined by BARC

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, MD, Study Chair — Fuwai central China cardiovascular hospotial
Locations (1):
- Fuwai central China cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No